CLINICAL TRIAL: NCT00003215
Title: Standard Chemotherapy (CHOP Regimen) Versus Sequential High-Dose Chemotherapy With Autologous Stem Cell Transplantation in Patients With Newly Diagnosed Aggressive Non-Hodgkin's Lymphomas and Poor Prognostic Factors: A Randomized Phase III Study (MISTRAL)
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Newly Diagnosed Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SAKK 38/97; SWS-SAKK-38/97; EU-97037
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic | interventions — Filgrastim; VAP-cyclo protocol; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Leucovorin; Melphalan; Methotrexate; Methylprednisolone; Mitoxantrone; Prednisone; Hydrocortisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: leucovorin calcium
Drug: melphalan
Drug: methotrexate
Drug: methylprednisolone
Drug: mitoxantrone hydrochloride
Drug: prednisone
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining peripheral stem cell transplantation with more than one drug regimen may kill more tumor cells. It is not known whether receiving standard combination chemotherapy alone is more effective than receiving multiple combination chemotherapy plus peripheral stem cell transplantation for aggressive non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is comparing giving different combination chemotherapy regimens together with peripheral stem cell transplantation to see how well they work in treating patients with newly diagnosed aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of sequential high-dose chemotherapy and autologous peripheral blood stem cell transplantation with standard chemotherapy (cyclophosphamide, doxorubicin, vincristine, and prednisone) in patients with newly diagnosed aggressive non-Hodgkin's lymphoma and poor prognostic factors.
* Compare the toxic effects of these 2 regimens in these patients.
* Compare the response rates and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive standard chemotherapy comprising cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP). Patients receive cyclophosphamide IV over 30 minutes, doxorubicin IV, and vincristine IV on day 1. Patients receive oral prednisone daily on days 1-5. Treatment repeats every 21 days for 6-8 courses. Patients with bulky disease at diagnosis or residual disease after chemotherapy receive radiotherapy 30-60 days after initiation of the last course of CHOP.
* Arm II: Patients receive 5 regimens of chemotherapy administered in sequence.

  * Regimen A : Patients receive CHOP as in Arm I.
  * Regimen B: Three weeks after starting regimen A, patients receive high-dose cyclophosphamide IV over 24 hours on day 1. Patients without initial bone marrow involvement receive filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 3 and continuing until autologous peripheral blood stem cells (PBSC) are harvested. PBSC are harvested on days 13-15 or when blood counts recover. Patients with initial bone marrow involvement do not undergo harvest of PBSC at this time, but receive G-CSF SC daily.
  * Regimen C: Two to three weeks after high-dose cyclophosphamide, patients receive vincristine IV and high-dose methotrexate IV over 6 hours on day 2. Patients receive leucovorin calcium IV every 6 hours on days 3-5 beginning 24 hours after initiation of the methotrexate infusion.
  * Regimen D: Within 1-2 weeks after the administration of methotrexate in regimen C, patients receive methylprednisolone IV followed 6 hours later by high-dose etoposide IV over 10 hours on day 1. Patients receive methylprednisolone IV on day 2. Patients without initial bone marrow involvement receive G-CSF SC daily beginning on day 3 and continuing until blood counts recover. Patients with initial bone marrow involvement receive G-CSF SC daily until autologous PBSC are harvested. PBSC are harvested on days 10-14 or when blood counts recover.
  * Regimen E: Myeloablative therapy and autologous PBSC transplantation begin 16-40 days after the administration of etoposide. Patients receive mitoxantrone IV over 1 hour every 2 hours for 3 doses on day 2 and melphalan IV over 30 minutes on day 5. PBSC are reinfused on day 6 beginning at least 24 hours after the administration of melphalan. Patients receive G-CSF SC or by continuous infusion beginning on day 7.

Patients with bulky disease at diagnosis or residual disease after chemotherapy receive radiotherapy 30-100 days after PBSC transplantation.

Patients at high risk of developing CNS disease receive prophylactic intrathecal chemotherapy. Patients may receive cytarabine, methotrexate, and hydrocortisone or methotrexate and hydrocortisone every 1-2 weeks for 6 courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 400 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma (NHL)

  * Diffuse large B-cell lymphoma
  * Primary mediastinal large B-cell lymphoma
  * Anaplastic large cell lymphoma (B-cell, T-cell, or null-cell type)
* At least two of the following risk factors:

  * Stage III or IV
  * LDH greater than upper limit of normal (ULN)
  * ECOG 2, 3, or 4
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 to 60

Performance status:

* See Disease Characteristics
* ECOG 0-4

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No hepatitis B or C
* AST or ALT no greater than 2 times ULN*
* Bilirubin no greater than 2.34 mg/dL* NOTE: *Unless due to tumor involvement

Renal:

* Creatinine clearance at least 60 mL/min (unless due to tumor involvement)

Cardiovascular:

* No significant heart failure
* LVEF normal
* No active angina pectoris
* No myocardial infarction within the past 6 months
* No major ventricular arrhythmia

Pulmonary:

* No significant lung disorder

Other:

* HIV negative
* No severe active acute or chronic infection
* No severe psychoses
* No prior or concurrent malignancy except adequately treated carcinoma in situ of the cervix or nonmelanomatous skin cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for NHL (except emergency therapy, but no more than 1 course of standard chemotherapy)

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for NHL (except emergency therapy of no greater than 600 cGy radiation)
* No concurrent prophylactic radiotherapy to the brain

Surgery:

* Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 1997-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Betticher, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (12):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Dr. Horst-Schmidt-Kliniken, Wiesbaden, Germany
- Saint Savvas Cancer Hospital of Athens, Athens, Greece
- European Institute of Oncology, Milan, Italy
- Switzerland (8):
  - Universitatsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital, Bern, Bern
  - Ratisches Kantons und Regionalspital, Chur
  - Hopital Cantonal Universitaire de Geneve, Collonge-Bellerive
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Result] Betticher DC, Martinelli G, Radford JA, Kaufmann M, Dyer MJ, Kaiser U, Aulitzky WE, Beck J, von Rohr A, Kovascovics T, Cogliatti SB, Cina S, Maibach R, Cerny T, Linch DC. Sequential high dose chemotherapy as initial treatment for aggressive sub-types of non-Hodgkin lymphoma: results of the international randomized phase III trial (MISTRAL). Ann Oncol. 2006 Oct;17(10):1546-52. doi: 10.1093/annonc/mdl153. Epub 2006 Aug 3. PMID 16888080